CLINICAL TRIAL: NCT02956772
Title: A Prospective Multicenter Randomized Controlled Open-label Trial of Transcatheter Arterial Chemoembolization (TACE) in Combination With Arsenic Trioxide Versus TACE in the Treatment of Middle-advanced Primary Hepatocellular Carcinoma (HCC) Patients
Brief Title: Transcatheter Arterial Chemoembolization (TACE) in Combination With Arsenic Trioxide Versus TACE in the Treatment of Middle-advanced Primary Hepatocellular Carcinoma (HCC) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hunan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xiang Hua, Dr., Hunan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RACE16001
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Primary Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TACE plus Arsenic Trioxide (Experimental): Patients in this group are to receive a single dose of TACE treatment on day 1, followed by arsenic trioxide at 10 mg/day for 14 days (day 8-21). TACE treatment is repeated every 9 weeks while arsenic trioxide every 3 weeks for treatment duration of 27 weeks. At least 3 cycles of arsenic trioxide are administrated.
  Interventions: Drug: TACE; Drug: Arsenic trioxide
- TACE (Active Comparator): Patients in this group are to receive a single dose of TACE treatment on day 1. TACE treatment is repeated every 9 weeks for 27 weeks.
  Interventions: Drug: TACE

INTERVENTIONS:
Drug: TACE — After the puncture of femoral artery via Seldinger method, a catheter was inserted and digital celiac axis or hepatic arteriography performed. Then a microcatheter was used to infuse chemotherapeutic agent (30 to 60 mg of pirarubicin) mixed with 5 to 20 mL of Lipiodol Ultra-Fluid. Embosphere microspheres (size of 100 to 300 um) were inserted for embolization.
Drug: Arsenic trioxide — Arsenic trioxide 10 mg is put into 500 ml saline solution and then administrated by continuous intravenous drip for 5 hours during a treatment day.
  Arms: TACE plus Arsenic Trioxide

SUMMARY:
A multicentre, randomized, open-label, parallel-group, active controlled study.

DETAILED DESCRIPTION:
Primary hepatocellular carcinoma (HCC) is one of the most common types of cancer and accounts for significant morbidity and mortality worldwide. Notably, more than half of the new HCC cases and deaths develop in China. Transarterial chemoembolization (TACE) has been proposed as the first-line therapeutic strategy for the treatment of patients with unresectable HCC. However, TACE has several limitations itself which might be potentially associated with tumor metastasis and relapse.

Recent studies have demonstrated that arsenic trioxide (As2O3) can act as the first-line therapeutic option in the treatment of acute promyelocytic leukemia. Thereafter, several small studies in China showed promising clinical benefits when As2O3 is administrated among the HCC patients. With these preliminary results, the investigators are planning to carry out a multicenter randomized controlled trial through which to explore the potential efficacy and safety of adjuvant As2O3 treatment for HCC patients.

ELIGIBILITY:
1. Subject is 18-80 years old.
2. Subject has no portal stem vein tumor thrombus.
3. Subject has primary middle-advanced liver cancer of Barcelona Clinic Liver Cancer stages B/C inappropriate for surgical resection or other locoregional therapy and still presents with tumor lesions in the liver.
4. Subject has evaluable tumor lesion(s) (using Magnetic Resonance Imaging /Computed Tomography) according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) Version 1.1: single lesion size ≥5cm or at least one lesion of >3cm in size when 2-3 lesions exist or there are 4 or more lesions.
5. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤1, Fibrosis index based on 4 factors (FIB-4)≤6 and an expected survival time of 12 weeks or more.
6. Haematology: white blood cell count ≥3.0×10^9/L; hemoglobin≥10 g/dL; blood platelet count≥80×10^9/L
7. Blood biochemistry: serum albumin ≥2.8 g/dL, total bilirubin ≤2 mg/dL or ≤34.2 umol/L, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 times of upper limit of normal (ULN); amylase and lipase ≤ 1.5 times of ULN; serum creatinine ≤2.0 mg/dL or < 1.5 times of ULN; estimated creatinine clearance ≥60 mL/min.
8. International normalized ratio (INR) is ≤ 2.3 or prothrombin time (PT) is ≤3 seconds than upper limit of normal control.
9. Echocardiogram indicated a left ventricular ejection fraction (LVEF) of >50%.
10. Subject has a liver function Child-Pugh class A or B.
11. Subject is not pregnant or lactating.
12. Female subjects must be infertile or agree to take effective contraceptives; male subjects and their partners of reproductive potential must also agree to use appropriate contraceptives.
13. Subject had no second tumor in the last 5 years, excluding skin basal cell carcinoma or skin squamous carcinoma or any other carcinoma in situ.
14. Subject had no history of systemic chemotherapy.
15. Subject has no any other concomitant anticancer therapies, such as local radiotherapy, systemic chemotherapy and molecular targeted therapy.
16. Subject and (or) guardian is able to understand this study and willing to provide written, informed consent to participate in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2-year
  Progression free survival (PFS) is defined as the time interval from the day of the random assignment to the first evidence of progression or death.

SECONDARY OUTCOMES:
Objective response rate | 2-year
  Tumor response is defined as complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to RECIST and will be assessed by the investigators. The tumor objective response rate (ORR) is calculated per treatment arm as the proportion of randomized patients having a confirmed best response of CR or PR.
Overall Survival | 2-year
  Overall survival will be measured from the date of randomization up to the date of death of any cause
Incidence of adverse events | Up to 2 years through study completion
  Toxicities will be evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v 4.0.

OTHER OUTCOMES:
Quality of life using EuroQol five dimensions five levels questionnaire | Baseline and week 6, 12, 18, 24 and 30 using EuroQol five dimensions five levels questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hua Xiang, Dr., Principal Investigator — Hunan Provincial People's Hospital
Locations (9):
- China (9):
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - Guizhou Province Tumor Hospital, Guiyang, Guizhou
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Xinjiang Medical University Cancer Hospital, Ürümqi, Xinjiang
  - The Tumor Hospital of Yunnan Province, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No